CLINICAL TRIAL: NCT02940613
Title: Do Visuals of Symptom Change Increase Rates of Rapid Response in First Weeks of CBT for Eating Disorders?
Brief Title: Using Visual Feedback to Influence Rapid Response in the Treatment of Eating Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, patients stopped attending treatment in person. Patients have not returned to in-person treatment, and there is no plan for this to occur. The study could not be conducted virtually in secure manner.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Michele Laliberte, Clinical Director and Psychologist, Eating Disorders Clinic, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STJOES2016PAC
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Bulimia Nervosa; Binge Eating Disorder
Keywords: Rapid response; Eating Disorders; Cognitive Behavior Therapy; Bulimia Nervosa; Binge Eating Disorder; Purging Disorder
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual feedback of symptom frequency (Experimental): Participants in this arm receive visual feedback of their symptom frequency over the first 4 weeks of active treatment, based on information they provide on a symptom checklist.
  Interventions: Behavioral: Visual feedback of symptom frequency
- No visual feedback of symptom frequency (No Intervention): Participants in this arm complete the symptom checklist as is typically done during treatment, but receive no visual feedback of their self-reported symptom frequency over the first 4 weeks of active treatment.

INTERVENTIONS:
Behavioral: Visual feedback of symptom frequency — Participants receive visual feedback of their symptom frequency over the first 4 weeks of active treatment, based on information they provide on a symptom checklist.
  Arms: Visual feedback of symptom frequency

SUMMARY:
This study has two aims: 1) to test the validity of an eating disorder symptom checklist against an established clinical interview; and 2) to examine whether providing eating disorder patients with visual graphs of their symptom frequency in the early sessions of active treatment will lead to higher numbers of patients achieving a "rapid response" (65% reduction in symptoms in the first 4 weeks of treatment). Groups where patients receive visual graphs of symptom frequency will be compared with groups where patients do not receive visual graphs of symptom frequency on rates of rapid response to cognitive behavior treatment for eating disorders.

DETAILED DESCRIPTION:
There is a growing body of research indicating that the best predictor of treatment outcome for eating disorders is a "rapid response" - or a 65% drop in symptoms such as binge eating or purging - in the first four weeks of Cognitive Behavior Treatment (CBT). Research is only now beginning to look at whether it is possible to increase the number of rapid responders by directly encouraging this behavior in patients. This study has two aims: 1) to validate information obtained about symptoms in a Weekly Symptom Checklist (WSC) against information obtained in clinical interview; and 2) to examine whether, in a context where rapid response is being discussed and actively encouraged, the rates of rapid response can be improved by providing patients with visual of symptom change in the first weeks of treatment. Investigators hypothesize that there will be significant correspondence between the WSC and clinical interview. Investigators also hypothesize that being given a visual of symptom change in the first weeks of treatment will result in higher rates of rapid response in patients being encouraged to achieve these objectives; and that rapid response will be related to higher rates of symptom remission at the end of treatment. Participants will be 40 patients diagnosed with Bulimia Nervosa, Binge Eating Disorder or Purging Disorder. These patients will be spread across 6 treatment groups. Three groups will be randomly selected (balanced across clinicians) to either receive or not receive visual feedback on change in frequency of symptoms based on their responses to the Weekly Symptom Checklist (WSC).

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index) over 19
* Diagnosis of Bulimia Nervosa, Binge Eating Disorder, or Other Specified Feeding and Eating Disorder (OSFED) Purging Disorder.

Exclusion Criteria:

* BMI below 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in eating disorder symptoms from baseline | Administered weekly up to week 25 (end of group treatment)
  Symptoms will be measured using a Weekly Symptom Checklist which asks participants to indicate frequency of the previous week's eating disorder symptoms (regular eating, objective and subjective binge eating, various methods of purging).

SECONDARY OUTCOMES:
The behavioral section of the Eating Disorders Examination (EDE) | At week 6, 10, and up to 25 weeks (end of group treatment)
  The behavioural section of the Eating Disorders Examination (EDE) will be modified to focus on the 28-day period directly prior to the assessment, rather than the prior 3 months as is typical. The behavioural section of the EDE assesses frequency of regular eating (i.e., meals and snacks) and frequency of eating disorder behaviours such as objective binge eating episodes, subjective binge eating episodes, frequency of self-induced vomiting, laxative use, diuretic use, and frequency and duration of exercise for compensatory or weight control purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Laliberte, Ph.D., Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
For reasons of confidentiality, only aggregated data will be made available.

REFERENCES:
- [Background] Agras WS, Crow SJ, Halmi KA, Mitchell JE, Wilson GT, Kraemer HC. Outcome predictors for the cognitive behavior treatment of bulimia nervosa: data from a multisite study. Am J Psychiatry. 2000 Aug;157(8):1302-8. doi: 10.1176/appi.ajp.157.8.1302. PMID 10910795
- [Background] Bulik CM, Sullivan PF, Carter FA, McIntosh VV, Joyce PR. Predictors of rapid and sustained response to cognitive-behavioral therapy for bulimia nervosa. Int J Eat Disord. 1999 Sep;26(2):137-44. doi: 10.1002/(sici)1098-108x(199909)26:23.0.co;2-n. PMID 10422602
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Fairburn CG, Agras WS, Walsh BT, Wilson GT, Stice E. Prediction of outcome in bulimia nervosa by early change in treatment. Am J Psychiatry. 2004 Dec;161(12):2322-4. doi: 10.1176/appi.ajp.161.12.2322. PMID 15569910
- [Background] Grilo CM, Masheb RM. Rapid response predicts binge eating and weight loss in binge eating disorder: findings from a controlled trial of orlistat with guided self-help cognitive behavioral therapy. Behav Res Ther. 2007 Nov;45(11):2537-50. doi: 10.1016/j.brat.2007.05.010. Epub 2007 Jun 7. PMID 17659254
- [Background] Grilo CM, Masheb RM, Wilson GT. Rapid response to treatment for binge eating disorder. J Consult Clin Psychol. 2006 Jun;74(3):602-13. doi: 10.1037/0022-006X.74.3.602. PMID 16822116
- [Background] Grilo CM, White MA, Wilson GT, Gueorguieva R, Masheb RM. Rapid response predicts 12-month post-treatment outcomes in binge-eating disorder: theoretical and clinical implications. Psychol Med. 2012 Apr;42(4):807-17. doi: 10.1017/S0033291711001875. Epub 2011 Sep 16. PMID 21923964
- [Background] Grilo CM, White MA, Masheb RM, Gueorguieva R. Predicting meaningful outcomes to medication and self-help treatments for binge-eating disorder in primary care: The significance of early rapid response. J Consult Clin Psychol. 2015 Apr;83(2):387-94. doi: 10.1037/a0038635. Epub 2015 Jan 26. PMID 25622201
- [Background] MacDonald DE, Trottier K, McFarlane T, Olmsted MP. Empirically defining rapid response to intensive treatment to maximize prognostic utility for bulimia nervosa and purging disorder. Behav Res Ther. 2015 May;68:48-53. doi: 10.1016/j.brat.2015.03.007. Epub 2015 Mar 17. PMID 25800137
- [Background] Masheb RM, Grilo CM. Rapid response predicts treatment outcomes in binge eating disorder: implications for stepped care. J Consult Clin Psychol. 2007 Aug;75(4):639-44. doi: 10.1037/0022-006X.75.4.639. PMID 17663617
- [Background] McFarlane TL, MacDonald DE, Royal S, Olmsted MP. Rapid and slow responders to eating disorder treatment: a comparison on clinically relevant variables. Int J Eat Disord. 2013 Sep;46(6):563-6. doi: 10.1002/eat.22136. Epub 2013 Apr 12. PMID 23580395
- [Background] McFarlane T, Olmsted MP, Trottier K. Timing and prediction of relapse in a transdiagnostic eating disorder sample. Int J Eat Disord. 2008 Nov;41(7):587-93. doi: 10.1002/eat.20550. PMID 18473336
- [Background] Olmsted MP, Kaplan AS, Rockert W, Jacobsen M. Rapid responders to intensive treatment of bulimia nervosa. Int J Eat Disord. 1996 Apr;19(3):279-85. doi: 10.1002/(SICI)1098-108X(199604)19:33.0.CO;2-J. PMID 8704727
- [Background] Olmsted MP, MacDonald DE, McFarlane T, Trottier K, Colton P. Predictors of rapid relapse in bulimia nervosa. Int J Eat Disord. 2015 Apr;48(3):337-40. doi: 10.1002/eat.22380. Epub 2014 Dec 26. PMID 25545720
- [Background] Raykos BC, Watson HJ, Fursland A, Byrne SM, Nathan P. Prognostic value of rapid response to enhanced cognitive behavioral therapy in a routine clinic sample of eating disorder outpatients. Int J Eat Disord. 2013 Dec;46(8):764-70. doi: 10.1002/eat.22169. Epub 2013 Aug 5. PMID 23913536
- [Background] Thompson-Brenner H, Shingleton RM, Sauer-Zavala S, Richards LK, Pratt EM. Multiple measures of rapid response as predictors of remission in cognitive behavior therapy for bulimia nervosa. Behav Res Ther. 2015 Jan;64:9-14. doi: 10.1016/j.brat.2014.11.004. Epub 2014 Nov 13. PMID 25462877
- [Background] Vall E, Wade TD. Predictors of treatment outcome in individuals with eating disorders: A systematic review and meta-analysis. Int J Eat Disord. 2016 Apr;49(4):432-3. doi: 10.1002/eat.22518. No abstract available. PMID 27084797
- [Background] Vaz AR, Conceicao E, Machado PP. Early response as a predictor of success in guided self-help treatment for bulimic disorders. Eur Eat Disord Rev. 2014 Jan;22(1):59-65. doi: 10.1002/erv.2262. Epub 2013 Oct 4. PMID 24123526
- [Background] Wilson GT, Fairburn CC, Agras WS, Walsh BT, Kraemer H. Cognitive-behavioral therapy for bulimia nervosa: time course and mechanisms of change. J Consult Clin Psychol. 2002 Apr;70(2):267-74. PMID 11952185
- [Background] Zunker C, Peterson CB, Cao L, Mitchell JE, Wonderlich SA, Crow S, Crosby RD. A receiver operator characteristics analysis of treatment outcome in binge eating disorder to identify patterns of rapid response. Behav Res Ther. 2010 Dec;48(12):1227-31. doi: 10.1016/j.brat.2010.08.007. Epub 2010 Sep 6. PMID 20869041